CLINICAL TRIAL: NCT03548805
Title: Randomized Controlled Study to Evaluate Safety and Efficacy of Ologen® Collagen Matrix Versus Mitomycin-C in Patients With Juvenile-onset Open Angle Glaucoma
Brief Title: Ologen® Collagen Matrix Versus Mitomycin-C in Patients With Juvenile-onset Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: Principal Investigator, HERF, Consultant-Ophthalmologist, L.V. Prasad Eye Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS-90616
Record Dates: First submitted 2018-03-16; First posted 2018-06-07 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy; Mitomycin

STUDY DESIGN:
Intervention Model Description: ologen® Collagen Matrix, Model 830601, shape Round cylindrical, Size 6mm (diameter) x 2mm (thickness),Manufacturer Aeon Astron Europe B. V.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trabeculectomy with Ologen (Experimental): ologen® Collagen Matrix
  Interventions: Procedure: ologen® Collagen Matrix
- Trabeculectomy with low dose mitomycin C (Active Comparator): Trabeculectomy with low dose MMC (0.02%)
  Interventions: Procedure: Trabeculectomy with low dose mitomycin C

INTERVENTIONS:
Procedure: ologen® Collagen Matrix — Ologen is a collagen matrix used to modulate wound healing in the postoperative period to promote diffuse blebs
  Arms: Trabeculectomy with Ologen
Procedure: Trabeculectomy with low dose mitomycin C — Trabeculectomy with low dose MMC
  Arms: Trabeculectomy with low dose mitomycin C

SUMMARY:
To the best of Investigator knowledge, no studies to this date have compared the safety and efficacyof ologen® Collagen Matrix to MMC in exaggerated healing response among JOAG patients. Given that,filtration surgery is usually less successful in patients with juvenile glaucoma; the purpose of this study is to compare these two adjuvant therapies in exaggerated healing response among JOAG patients. Investigator hypothesis is that trabeculectomy with ologen® Collagen Matrix would be as effective as MMC in IOP control, with prominent bleb morphology as compared to MMC bleb.

DETAILED DESCRIPTION:
Standard trabeculectomy All trabeculectomy surgeries will be performed under peribulbar anesthesia.Under aseptic surgical technique, superior rectus suture will be placed using 4-0 silk and a fornix-based conjunctival flap will be performed. Sub-Tenon dissection and hemostasis may be performed as required.A half-thickness 4 x 4mm rectangular/ triangular scleral flap will be dissected up to clear cornea, and a 2 × 2 mm deep scleral block will be excised and peripheral iridectomy will be performed. The scleral flap will be closed with one or two 10-0 nylon sutures and conjunctiva will be closed with 8-0 vicryl suture. Releasable sutures may be applied to the scleral flap if needed.

ologen® Collagen Matrix ologen® Collagen Matrix approved by Indian health authority with registration numberof MD-1517 (valid till Mar-15-2018) will be provided by Aeon Ajanta India Pvt. Ltd. free of cost for this clinical research only.

The following table summarizes the model number, shape and manufacturer of ologen® Collagen Matrix to be used in this clinical research.

Product Model Shape Size Manufacturer Country of Origin Product Registration ologen® Collagen Matrix 830601 Round cylindrical 6mm (diameter) x 2mm (thickness) Aeon Astron Europe B. V. The Netherlands MD-1517 (valid till Mar-15-2018)

Mitomycin C Mitomycin-C Kyowa®; Kyowa Hakko Kogyo Co., Ltd. will be used. 0.02% solution of MMC will be prepared freshly on the day of planned surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 10 to 40 years (inclusive)
2. Uncontrolled IOP (defined as IOP > 21 mm Hg) despite maximum tolerable antiglaucoma therapy
3. Open anterior chamber angle on gonioscopic examination
4. Glaucomatous optic disc damage on clinical examination (focal or diffuse neuroretinal rim thinning, localized notching or nerve fiber layer defects) with corresponding visual field (VF) defects
5. Patientor his/her guardian is willing and able to comply with study procedures and sign informed consent

Exclusion Criteria:

1. Patients with steroid-induced glaucoma and other types of secondary open angle glaucoma 2. Juvenile-onset Open Angle Glaucoma eyes that underwent trabeculectomy with MMC or had a previous filtering surgery 3. Patients with any other ocular disease that may expose them to an undue risk of a significant adverse event during the course of the study, including but not limited to ocular cancer, trauma, corneal surface damage or other conditions as determined by the clinical judgment of the investigator 4. Patient with single functional eye 5. Participation in any study 30 days prior to trabeculectomy 6. Pregnant or breast-feeding women

-

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure control in the two groups will be compared. | 1 year
  Comparison of IOP control between the two groups: Assess control of IOP over time. "Complete success" is defined as IOP reduction of >20% and / or an IOP constantly <21 mmHg without any antiglaucoma medication. "Qualified success" is defined as IOP < 21 mmHg with topical antiglaucoma medication. "Failure" is defined as IOP > 21mmHg in 2 subsequent follow visits despite topical antiglaucoma medication.

SECONDARY OUTCOMES:
Bleb morphology:Change of Moorfields Bleb Grading System (MBGS) score over time | at 3 months, 6 months and 1 year
  Assess bleb characteristics using Moorfields Bleb Grading System (MBGS) score as measurement tool to document bleb grading score over time; and comparison of bleb morphology in the two groups with photographs and ASOCT

CONTACTS AND LOCATIONS:
Overall Officials: Senthil Sirisha, MS, Principal Investigator — YES
Locations (1):
- L V Prasad Eye Institute, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No